CLINICAL TRIAL: NCT02567344
Title: A Double Blind, Sham Controlled Trial of Excitatory rTMS to the Left Dorsolateral Pre-Frontal Cortex to Reduce Cannabis-Cue Induced Craving and Impulsive Decision Making in Cannabis Use Disordered Participants.
Brief Title: Excitatory rTMS to the Left Dorsolateral Pre-Frontal Cortex to Reduce Cannabis-Cue Induced Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00047358
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-05

CONDITIONS: Cannabis
Keywords: Cannabis; rTMS; Craving; Decision making
MeSH Terms: conditions — Marijuana Abuse | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Experimental): Active rTMS will be delivered to the Left DLPFC at 10Hz. A total of 4000 pulses will be delivered.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): Sham rTMS will be delivered to the Left DLPFC at 10 Hz using an electronic sham system used in multiple other investigations. A total of 4000 pulses of sham rTMS will be delivered.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS will be delivered at 110% rMT to the Left DLPFC with 5 seconds on, 10 seconds off for 4000 pulses.
  Arms: Active rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation — rTMS will be delivered via an electronic sham coil that mimics real rTMS in appearance, sound, and feeling. Pulses will be delivered to the Left DLPFC with 5 seconds on, 10 seconds off for 4000 pulses.
  Arms: Sham rTMS

SUMMARY:
This is a double-blind, crossover trial that will recruit a cohort of non-treatment seeking Cannabis use disordered participants. Participants will then undergo either active, or sham rTMS to the LDLPFC, and cue-induced craving, and risky decision making will be assessed.

DETAILED DESCRIPTION:
Our primary aims are to determine the effect of a single session of 10 Hz L DLPFC rTMS on cannabis cue induced craving (Aim1), and behavioral tasks of impulsive decision making (Aim2), in non-treatment seeking individuals with Cannabis Use Disorder. The aims of the study will be accomplished by performing a double-blind, sham-controlled crossover trial. Non-Treatment seeking individuals with CUD will be recruited through media advertisements, as well as via a pre-established database of non-treatment seeking individuals who have participated in previous Cannabis trials and agreed to be re-contacted. Interested individuals will undergo a brief phone screen to determine if they meet general inclusion/exclusion criteria, and if so will be invited to meet with study personnel in order to sign informed consent, and undergo a screening visit. There will then be two experimental visits separated by at least one week. During each of these visits participants will undergo either a real, or sham rTMS treatment, as well as a cannabis cue Paradigm. Data on craving as well as on impulsive decision making will be collected before and after each treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Participants must be between the ages of 18 and 60.
3. Participants must meet DSM-V criteria for Cannabis Use Disorder, with use of at least 20 days/month.
4. Participants must agree to abstinence from Cannabis for at least 24 hours prior to each visit.
5. Participants must have a Positive UDS for cannabis (confirming they are regular users), and a negative salivary cannabis test (Confirming no use within 10-14 hours)

Exclusion Criteria:

1. Participants must not be pregnant and participate in the study.
2. Participants must not test positive for any substance other than cannabis on UDS.
3. Participants must not meet criteria for any other Substance Use Disorders with the exception of Nicotine Use Disorder.
4. Participants must not be on any medications that have central nervous system effects.
5. Participants Must not have a history of/or current Psychotic disorder.
6. Participants must not have a history of Dementia or other cognitive impairment.
7. Participants must not have active suicidal ideation, or suicide attempt within the past 90 days.
8. Participants must not have any contraindications to receiving rTMS as assessed by the TMS safety sheet.
9. Participants must not have any unstable general medical conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Marijuana Craving Questionnaire (MCQ) | 15 Minutes
  The MCQ will be given before and after a marijuana-cue paradigm, and the primary outcome will be the change score from pre to post.

SECONDARY OUTCOMES:
The Balloon Aptitude Response Task (BART) | 30 Minutes
  The BART will be given pre, and post rTMS. Number of corrected pumps, and number of burst balloons will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — MUSC department of psychiatry